CLINICAL TRIAL: NCT05728255
Title: Assessment of the Mechanism of Non-cardiac Syncope by 24-hour Ambulatory Blood Pressure Monitoring (ABPM) and Tilt-table Short Cardiovascular Autonomic Function Battery (SCAFB)
Brief Title: Assessment of the Mechanism of Non-cardiac Syncope
Acronym: 2STEPS
Status: Completed | Type: Observational
Sponsor: Istituto Auxologico Italiano (Other)
Responsible Party: Sponsor
Other Study IDs: 09C337
Record Dates: First submitted 2023-02-04; First posted 2023-02-15 (Actual); Last update posted 2024-07-17 (Actual); Status verified 2024-07

CONDITIONS: Syncope; Syncope, Vasovagal; Orthostatic Hypotension; Syncope, Carotid Sinus
Keywords: Syncope; Orthostatic hypotension; Tilt table test; Ambulatory blood pressure monitoring
MeSH Terms: conditions — Syncope; Syncope, Vasovagal; Hypotension, Orthostatic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: ABPM plys SCAFB — 24-hour ambulatory blood pressure monitoring (ABPM) and of tilt-table Short Cardiovascular Autonomic Function Battery (SCAFB) which consists in carotid sinus massage (CSM) and head-up tilt test (HUT) performed one after the other in an uninterrupted sequence as a single procedure on a tilt table

SUMMARY:
Identifying the mechanism of non-cardiac syncope is the essential prerequisite for an effective personalized therapy.

Aim of this multicentre, prospective, cross-sectional, observational study is to assess effectiveness and diagnostic yield of a two-step standardized assessment which consists of 24-hour ambulatory blood pressure monitoring (ABPM) and of tilt-table Short Cardiovascular Autonomic Function Battery (SCAFB) which consists in carotid sinus massage (CSM), limited to patients ≥40-year-old, standing test, and head-up tilt test (HUT) performed one after the other in an uninterrupted sequence as a single procedure on a tilt table

DETAILED DESCRIPTION:
Identifying the mechanism of non-cardiac syncope is the essential prerequisite for an effective personalized therapy. Indeed, the choice of appropriate therapy and its efficacy are largely determined by the mechanism of syncope rather than its aetiology or clinical presentation. The identified mechanism of syncope should be carefully assessed and assigned either to hypotensive or bradycardic phenotype, which will determine the choice of therapy (counteracting hypotension or counteracting bradycardia).

Several tests have been developed to identify the mechanism of non-cardiac syncope. The great number of tests, most of them being time-consuming, is one of the barriers for widespread utilization in the busy clinical practice. They are expensive and often not fully reimbursed by the health services.

Aim of this multicentre, prospective, cross-sectional, observational study is to assess effectiveness and diagnostic yield of a two-step standardized assessment which consists of 24-hour ambulatory blood pressure monitoring (ABPM) and of tilt-table Short Cardiovascular Autonomic Function Battery (SCAFB). SCAFB consists in carotid sinus massage (CSM), limited to patients ≥40-year-old, standing test, and head-up tilt test (HUT) performed one after the other in an uninterrupted sequence as a single procedure on a tilt table

The study hypothesis is that these two investigations, performed in sequence, can identify the mechanism of syncope in most of the patients in a quick and easy-to-perform way and at relatively low costs.

ELIGIBILITY:
Inclusion Criteria:

* severe recurrent non-cardiac syncope referred for assessment of the mechanism of syncope. Non-cardiac syncope is diagnosed when the clinical features are consistent with reflex syncope and orthostatic hypotension, and cardiac syncope is ruled out .

Exclusion Criteria:

1. Non-syncopal causes of real or apparent loss of consciousness that may be incorrectly diagnosed as syncope (eg, unexplained falls, epilepsy, psychogenic pseudosyncope and other rare causes)
2. Established or suspected cardiac syncope in complying with the criteria of the European Society of Cardiology (ESC) syncope guidelines (1). Specifically, these were the patients with: (i) suspected cardiac arrhythmic syncope [inadequate sinus bradycardia (<50 b.p.m.) or sinoatrial block, second-degree Mobitz I atrioventricular block, second-degree Mobitz II or third-degree atrioventricular block, paroxysmal tachyarrhythmia or ventricular tachycardia, bundle branch block]; (ii) severe structural heart disease and/or significant ECG abnormalities, as defined in Table 2 of those guidelines (1).
3. Classical orthostatic hypotension diagnosed at the initial evaluation by Active Standing test
4. Constitutional or drug-induced persistent hypotension already diagnosed at the initial evaluation by office BP measurement or previous historical features
5. Non-severe forms of non-cardiac syncope, i.e., patients with rare and mild episodes occurring in low-risk situations. In these patients the investigation of the underlying mechanism of syncope is not necessary and treatment strategies are mainly based on education on preventive measures, lifestyle modification, and reassurance regarding the benign nature of the condition.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with severe syncopes are those patients who are asking for mechanism-specific therapy because they are affected by recurrent syncopes impairing quality of life or have syncopes with absent or very short prodrome increasing the risk of injuries or are at risk of syncope during high-risk activities (e.g., driving, machine operation, flying, or competitive athletics, etc.).
Sampling Method: Probability Sample
Enrollment: 330 (Actual)
Dates: Start 2024-04-01 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
Prevalence | 1 month
  Prevalence of hypotensive and bradycardic phenotypes

SECONDARY OUTCOMES:
Diagnostic yield | 1 month
  Diagnostic yield of ABPM and of SCAFB
Diagnosis | 1 month
  Case mix of etiologic diagnoses

CONTACTS AND LOCATIONS:
Locations (8):
- University of marseille Aix en Provence, Marseille, France
- Italy (4):
  - IRCCS Istituto Auxologico Italiano, Milan, MI
  - University of Florence, Florence
  - ospdali del Tigullio, Lavagna
  - Università della Campania Vamvitelli, Naples
- AMC Universisty of Amsterdam, Amsterdam, Netherlands
- University of Barcelona Vall d'Ebron, Barcelona, Spain
- Karolinska Institut, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rivasi G, Groppelli A, Brignole M, Soranna D, Zambon A, Bilo G, Pengo M, Sharad B, Hamrefors V, Rafanelli M, Testa GD, Rice C, Kenny RA, Sutton R, Ungar A, Fedorowski A, Parati G. Association between hypotension during 24 h ambulatory blood pressure monitoring and reflex syncope: the SynABPM 1 study. Eur Heart J. 2022 Oct 11;43(38):3765-3776. doi: 10.1093/eurheartj/ehac347. PMID 35766175
- [Result] Brignole M, Rivasi G. New insights in diagnostics and therapies in syncope: a novel approach to non-cardiac syncope. Heart. 2021 Jun;107(11):864-873. doi: 10.1136/heartjnl-2020-318261. Epub 2021 Jan 18. PMID 33462120